CLINICAL TRIAL: NCT05187793
Title: A Multicenter, Open-label, Randomized Study of the Efficacy and Safety of Artlegia (INN: Olokizumab) New Dosing Regimen in Patients With Coronavirus Infection (COVID-19) With Signs of Hyperinflammation
Brief Title: Study of Efficacy of Different Treatment Regimens of Olokizumab
Acronym: RESET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: R-Pharm (Industry)
Collaborators: Federal Budget Institution of Science "Central Research Institute of Epidemiology" of the Rospotrebnadzor (Unknown); Group of companies Medsi, JSС (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL04041094
Record Dates: First submitted 2021-12-24; First posted 2022-01-12 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; 2019-nCoV; Severe acute respiratory syndrome coronavirus 2
MeSH Terms: conditions — COVID-19 | interventions — olokizumab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olokizumab (Experimental): Subject randomized to receive intravenous infusion of 0,8 ml solution of Olokizumab, one (128 mg), or two (256 mg) doses, in addition to standard therapy in line with the current temporary guidelines "Prevention, diagnosis and treatment of new coronavirus infection (COVID-19)" of the Ministry of Health of Russian Federation.
  Standard therapy includes:
  * Baricitinib, p.o., 4 mg once daily for 7 days
  * Favipiravir, p.o.,
    * for patients weighing <75 kg: 1600 mg twice daily on Day 1, then 600 mg twice daily from the 2nd to the 10th day;
    * for patients weighing ≥ 75 kg: 1800 mg twice daily on Day 1, then 800 mg twice daily from the 2nd to the 10th day; (Patients who have started etiotropic therapy with favipiravir or remdesivir prior to randomization will continue the initiated treatment.)
  * dexamethasone at doses of 4 - 20 mg / day or methylprednisolone at a dose of 1 mg / kg / intravenous injection every 12 hours.
  Interventions: Drug: Olokizumab; Drug: Standard therapy
- Standard therapy (Active Comparator): Standard therapy in line with the current temporary guidelines "Prevention, diagnosis and treatment of new coronavirus infection (COVID-19)" of the Ministry of Health of Russian Federation including:
  * Baricitinib, p.o., 4 mg once daily for 7 days
  * Favipiravir, p.o.,
    * for patients weighing <75 kg: 1600 mg twice daily on Day 1, then 600 mg twice daily from the 2nd to the 10th day;
    * for patients weighing ≥ 75 kg: 1800 mg twice daily on Day 1, then 800 mg twice daily from the 2nd to the 10th day; (Patients who have started etiotropic therapy with favipiravir or remdesivir prior to randomization will continue the initiated treatment.)
  * dexamethasone at doses of 4 - 20 mg / day or methylprednisolone at a dose of 1 mg / kg / intravenous injection every 12 hours.
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: Olokizumab — Olokizumab, 128 mg, solution for subcutaneous administration 160 mg/mL
  Arms: Olokizumab
Drug: Standard therapy — Standard treatment including:
  * Baricitinib, 4 mg, film coated tablets
  * Favipiravir, 200 mg, film coated tablets
  * Dexamethasone IV or IM OR Methylprednisolone IV

SUMMARY:
The primary objective of the study is to evaluate the efficacy and safety of Artlegia (INN: olokizumab) new dosing regimen in patients with moderate coronavirus infection (COVID-19) with signs of hyperinflammation.

This study is a multicentre, open-label, randomized, comparative, parallel group, active-controlled clinical trial.

DETAILED DESCRIPTION:
The study has an adaptive design. According to the initial calculation of the sample size it was planned to include about 204 patients in the study. After interim analyzing of the data of the first 100 randomized patients a decision about the final sample size was made. The size of the intent-to-treat (ITT) population for the final efficacy analysis at the primary endpoint is 180 patients. Taking into account the probability of dropping out up to 10% of patients, 198 patients were planned to be randomized into the study, no more than 220 patients were planned to be screened.

The study will include the following periods:

* Screening period lasting up to 2 days (days -1-0). During this period patient's eligibility assessment will be performed;
* Treatment period: up to 10 days. Treatment period starts from the end of the screening (days 1-10) and includes randomization following by a 10 days of standard therapy with or without olokizumab and patient monitoring (laboratory tests, electrocardiogram (ECG), chest computed tomography (CT));
* Short-term follow-up period up to 28 days (days 11 through 28). It includes procedures of patient monitoring (laboratory tests, ECG, chest CT) on days 14 (± 2) and 28 (± 2).
* Long-term follow-up period: up to 180 days (days 29 through 180). Includes telephone contacts with the patient on days 45, 60, 90 and 180.

Eligible patients will be randomized to one of 2 treatment groups to receive olokizumab (OKZ) 128 mg i.v. infusion (one or two single doses) against the background of standard therapy, or standard therapy alone.

In OKZ group study drug olokizumab 128 mg is administered as a single intravenous infusion. A comprehensive assessment of the clinical and laboratory response is performed daily within 5 days (120 hours) after the first injection. If there is no response to therapy or the response is insufficient, the repeated dose of OKZ, 128 mg, is administered.

As standard anti-inflammatory therapy, patients in both groups will receive baricitinib (at the standard recommended dose of 4 mg / 1 time per day, for 7 days) and low doses of glucocorticosteroids (dexamethasone at doses of 4-20 mg / day or methylprednisolone at a dose of 1 mg / kg / intravenous injection every 12 hours).

With an observed clinical deterioration (fever increase, dyspnea, oxygen saturation decrease, the appearance / increase in the need for oxygen support) after repeated infusion of OKZ in the main group (at least 24 hours from the first infusion started), or after 24 hours or more from the start of therapy in the comparison group, the patient is considered "not responding" to therapy and requiring another anti-inflammatory treatment regimens.

Standard therapy also includes etiotropic therapy for COVID-19, as well as symptomatic and anticoagulant therapy.

Etiotropic therapy. Favipiravir will be used in recommended dosage regimens according to temporary guidelines "Prevention, diagnosis and treatment of new coronavirus infection (COVID-19)" of the Ministry of Health of Russian Federation.

Patients who have started etiotropic therapy with favipiravir or remdesivir prior to randomization will continue the initiated treatment.

Сlinical status will be assessed daily in the first 10 days, then on days 14, 21, 28, 45, 60, 90 and 180, vital signs - three times daily in the first 5 days, once daily on days 6-10, then on days 14 and 28, chest CT - on days 7, 14 and 28; laboratory parameters - on days 1 - 5, 10, 14, 28.

On day 7 primary endpoint of patient's clinical recovery (defined as score of 3 or less on a 10-point ordinal scale of clinical improvement) will be assessed. The last patient's visit to the study site will be the visit on Day 28. On Days 45, 60, 90 and 180 the phone follow-up will be performed.

In olokizumab group, eligible subjects will be selected to participate in pharmacokinetic analysis. Blood samples for the evaluation of olokizumab pharmacokinetics will be taken before the infusion of olokizumab and in 2 h, 4 h, 8 h, 24 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 h, 192 h, 216 h, 240 h, 336 h and 672 h after the first administration of the drug (since the start of infusion).

Expected study duration for each patient will be 182 (± 2) days, including screening periods (2 days), therapy and short-term follow-up (28 (± 2) days), and long-term extended follow-up (152 (± 2) 2 days).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent for participation in this study.
2. Hospitalization (no more than 72 hours prior to randomization) with a diagnosis of coronavirus infection caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) virus (COVID-19).
3. Moderate COVID-19. Moderate course of the disease is characterized by pneumonia on chest computed tomography (CT) (CT-1,2 stages) and body temperature > 38 °C, in combination with 1 or more of the following:

   * SpO2 <95%,
   * respiratory rate > 22,
   * dyspnea on exertion,
   * C-reactive protein (CRP) level> 10 mg / l,
   * one of the following risk factors: diabetes mellitus, severe cardiovascular disease, chronic renal failure, cancer, obesity, or age ≥ 65 years.
4. The presence of signs of hyperinflammation. Signs of hyperinflammation are body temperature ≥ 38 °C for 2 days or more, combined with 1 or more of the following:

   * CRP level > 3 Upper Normal Limit (UNL),
   * White blood cell count - 2.0-3.5 × 10^9 / l,
   * Absolute lymphocyte count - 1.0-1.5 × 10^9 / l
5. Infection caused by the SARS-CoV-2 confirmed by of Polymerase chain reaction (PCR) test or an express test for antigen / antibodies to SARS-CoV-2 framework of the protocol.
6. Ability to follow protocol requirements and perform all clinical trial procedures.
7. The willingness of the participants and their sexual partners to use reliable methods of contraception, during the entire study and at least 3 months after the treatment completion. This requirement does not apply to participants who have undergone surgical sterilization as well as to women with permanent cessation of menstruation, which should be determined retrospectively after 12 months of natural amenorrhea, i.e. amenorrhea with an appropriate clinical status (eg, appropriate age). Reliable methods of contraception involve the use of one barrier method in combination with one of the following: spermicides, intrauterine spiral/oral contraceptives in a sexual partner.
8. Willingness not to drink alcohol during the entire study.

Additional inclusion criteria for the pharmacokinetics (PK) subgroup:

1. Signed informed consent to participate in the additional study of pharmacokinetics.
2. Body mass index 18.5 - 35.0 kg/m2.
3. The ability of the patient, by the opinion of the investigator, to participate in the additional study of pharmacokinetics and to provide the required number of blood samples.

Exclusion Criteria:

1. Hypersensitivity to olokizumab and / or other components of the study drug.
2. Contraindications to favipiravir or glucocorticosteroids or Janus kinase inhibitors (baricitinib).
3. Signs of a severe or extremely severe course of COVID-19, such as:

   * altered level of consciousness, agitation,
   * the need for / use of Non-invasive ventilation (NIV) / Adaptive lung ventilation (ALV) / Extracorporeal membrane oxygenation (ECMO) at screening,
   * hemodynamic instability eg systolic blood pressure < 90 mm Hg or diastolic blood pressure < 60 mm Hg and urine output less than 20 ml / hour,
   * CT-3,4 stage on chest CT, signs of Acute respiratory distress syndrome (ARDS),
   * arterial blood lactate > 2 mmol / l,
   * quick Sequential Organ Failure Assessment (qSOFA) > 2 points.
4. Any of the following laboratory abnormalities:

   * Hemoglobin <80 g / l,
   * Absolute neutrophil count <0.5 x 10^9 / l,
   * White blood cell count <2.0 x 10^9 / l,
   * Platelet count <50 x 10^9 / l,
   * Alanine transaminase (ALT) and / or Aspartate aminotransferase (AST) ≥ 3.0 x UNL.
5. Severe renal failure: creatinine clearance < 30 ml / min.
6. Confirmed sepsis with non-COVID-19 pathogens and procalcitonin levels > 0.5 ng / ml.
7. Prior hepatitis B and / or C virus infection.
8. High probability of disease progression to death within the next 24 hours, regardless of therapy, by the opinion of the investigator.
9. Concomitant diseases associated with a poor prognosis (with the exception of those listed in inclusion criteria No. 3: diabetes mellitus, severe cardiovascular disease, chronic renal failure, cancer, obesity, or age ≥ 65 years).
10. Immunosuppressive therapy for organ transplantation.
11. Recent (less than 5 half-lives) or prescribed at screening:

    * Olokizumab (use or prescription prior to study randomization);
    * Biological drugs with immunosuppressive effects, including, but not limited to:Interleukin 1 (IL-1) inhibitors (anakinra, canakinumab), IL-6 receptor inhibitors (tocilizumab, sarilumab, levilimab), IL-17 (secukinumab, netakimab), tumor necrosis factor α inhibitors (TNFα) (infliximab, adalimumab, etanercept, etc.), anti-B-cell drugs, and others;
    * Immunosuppressive drugs (including, but not limited to):

      * glucocorticoids in high doses (> 1 mg / kg prednisolone equivalent) orally or parenterally;
      * Janus kinase (JAK) kinase inhibitors;
      * cyclophosphamide, etc.
12. History of active tuberculosis or suspected active tuberculosis.
13. Simultaneous participation in another clinical trial.
14. Pregnancy or breastfeeding at screening; planning pregnancy during the entire study and within 3 months after the completion of treatment.
15. Any information from anamnesis that may lead to a complicated interpretation of the study results or create additional risk for the patient as a result of participation in the study.
16. Known (from history) or suspected abuse of alcohol, psychotropic drugs; drug addiction.
17. Subjects with a history or presence of any psychiatric disorder(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Clinical recovery rate at day 7 | Up to day 7
  Clinical recovery defined as score of 3 or less on a 10-point ordinal scale of clinical improvement.
  (From 0 "Healthy - no clinical manifestations, no viral RNA detected" to 10 "Death".) 7 days are counted from the day of the first administration / intake of study therapy / comparison therapy, depending on study group.
  Criteria for transition from category "4" to category "3" (criteria for potential discharge): body temperature < 37 °C; respiratory rate ≤ 20 per minute; SpO2 ≥ 95% without oxygen support, CRP < 10 mg/l. If any emergency procedures should be prescribed and/or signs of progression on CT are detected, the patient cannot be discharged/transferred to category "3".
  (In the case of the "rescue" therapy use or the development of clinical deterioration (an increase in the score by 1 point or more) during the follow-up period in a previously recovered patient, the patient is not considered as a "responder", i.e., who has reached the primary endpoint.)

SECONDARY OUTCOMES:
Rate of clinical deterioration by at least 1 point from the baseline ordinal score at day 28, depending on study group | Up to day 28
  Rate of clinical deterioration by at least 1 point from the baseline ordinal score at day 28, depending on study group
CRP normalization rate | Up to Day 28
  Normalization is defined as CRP blood level within normal range (< 10 mg/l), assessed on days 5, 10, 14, 28, depending on study group.
Ferritin normalization rate | Up to Day 28
  Normalization is defined as ferritin blood level within normal range, assessed on days 5, 10, 14, 28, depending on study group.
D-dimer normalization rate | Up to Day 28
  Normalization is defined as D-dimer blood level within normal range, assessed on days 5, 10, 14, 28, depending on study group.
Mean CRP levels | Up to Day 28
  Mean CRP levels assessed on days 5, 10, 14, 28, depending on study group
Mean ferritin levels | Up to Day 28
  Mean ferritin levels assessed on days 5, 10, 14, 28, depending on study group
Mean D-dimer levels | Up to Day 28
  Mean D-dimer levels assessed on days 5, 10, 14, 28, depending on study group
Rate of prescribing other anti-inflammatory therapy regimens (rescue therapy), depending on study group | Up to day 28
  Rate of prescribing other anti-inflammatory therapy regimens (rescue therapy), depending on study group

OTHER OUTCOMES:
Rate of clinical deterioration by at least 1 point from the baseline ordinal score at day 7, depending on study group | Up to day 7
  Rate of clinical deterioration by at least 1 point from the baseline ordinal score at day 7, depending on study group
Clinical recovery rate at day 14 | Up to day 14
  Clinical recovery defined as score of 3 or less on a 10-point ordinal scale of clinical improvement, 14 days are counted from the day of the first administration / intake of study / comparison therapy by treatment group
Cumulative incidence of transfer to intensive care unit (ICU), transfer to mechanical ventilation, development of ARDS and / or death, at day 28 | Uo to day 28
  Cumulative incidence of transfer to ICU, transfer to mechanical ventilation, development of ARDS and / or death, at day 28
Incidence of progression on chest CT at day 28 | Up to day 28
  Incidence of progression on chest CT at day 28, depending on study group
Rate of transfer to ICU at day 28 | Up to day 28
  Rate of transfer to ICU at day 28, depending on study group
Rate of transfer to mechanical ventilation at day 28 | Up to day 28
  Rate of transfer to mechanical ventilation at day 28, depending on study group
Incidence of ARDS at day 28 | Up to day 28
  Incidence of ARDS at day 28, depending on study group
Incidence of death from any cause at day 28 | Up to day 28
  Incidence of death from any cause at day 28, depending on study group
Incidence of symptoms of a secondary bacterial infection | Up to day 28
  * leukocytosis > 12x10^9 / l (in the absence of previous use of glucocorticosteroids),
  * and / or shift to stab > 10 %,
  * and / or purulent sputum or other clinical manifestations of purulent inflammation,
  * and / or an increase in procalcitonin> 0.5 ng / ml depending on study group
Time to improvement in clinical status by at least 1 point | from the moment of drug administration to improvement, up to 28 days
  Time to improvement in clinical status by at least 1 point (from the moment of drug administration) (median, in days), depending on study group
Incidence of improvement in clinical status by at least 1 point on days 3, 5, 7, 10, 14, 21, 28, depending on study group | Up to day 28
  Incidence of improvement in clinical status by at least 1 point on days 3, 5, 7, 10, 14, 21, 28, depending on study group
Time to reach SpO2 ≥ 95%, without oxygen support for 2 consecutive days | from the moment of drug administration to the moment when SpO2 ≥ 95%, up to 28 days
  Time to reach SpO2 ≥ 95%, without oxygen support for 2 consecutive days (from the moment of drug administration) (median, in days), depending on study group
Duration of hospitalization at day 28 | from the moment of drug administration to discharge, up to 28 days
  Duration of hospitalization at day 28 (from the moment of drug administration) (median, in days), depending on study group
Duration of ICU stay at day 28 | from the moment of drug administration to discharge from ICU, up to 28 days
  Duration of ICU stay at day 28 (from the moment of drug administration) (median, in days), depending on study group
Time to normalization of temperature | from the moment of drug administration to temperature normalization, up to 28 days
  Time to normalization of temperature (body temperature less than 37 °C for 48 hours or more, without taking antipyretics) (from the moment of drug administration) (median, in days), depending on study group
Change from baseline of the assessment of the immune status by the Investigator | Baseline, day 28
  Change from baseline of the assessment of the immune status by the Investigator, based on clinical course and laboratory markers (- IL-6, - complement components - C3 and C4, T-lymphocytes (CD3 + CD19-); T - helpers (CD3 + CD4 + ); T - cytotoxic lymphocytes (CD3 + CD8); Immunoregulatory index (T-helpers / T-cytotoxic), (CD3 + CD4 + / CD3 + CD8 +); B - lymphocytes (CD3-CD19 +); Activated T-lymphocytes with phenotype (CD3 + HLA-DR +); Lymphocytes with HLA-DR + phenotype, NK cells total (CD3- CD16 + CD56 +); Activated T-cells with markers of NK cells (CD3 + CD56 +).

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (5):
- Russia (5):
  - State Budgetary Healthcare Institution "City Clinical Hospital named after F.I. Inozemtsev of Moscow Healthcare Department", Moscow
  - Federal State Budgetary Institution "Central Clinical Hospital with a Polyclinic" of Presidential Administration of the Russian Federation, Moscow
  - State Budgetary Healthcare Institution "City Clinical Hospital № 52 of Moscow Healthcare Department", Moscow
  - State Budgetary Healthcare Institution "Infectious Diseases Hospital No. 1 of Moscow Healthcare Department", Moscow
  - State Budgetary healthcare Institution of the Voronezh region "Voronezh Regional Clinical Hospital No. 1", Voronezh

IPD SHARING:
Plan to Share IPD: No